CLINICAL TRIAL: NCT01887470
Title: A Randomized, Single-blind Pilot Study to Determine the Safety, Efficacy, and Patient Preference of 2 Regimens of Lactulose for Cleansing of the Colon as a Preparation for Colonoscopy in Adults
Brief Title: 2 Regimens of Lactulose for Colonoscopy Preparation in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CPI-KR-004
Record Dates: First submitted 2013-06-21; First posted 2013-06-26 (Estimated); Results first posted 2015-06-01 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Colonoscopy Preparation
Keywords: Bowel Evacuation; Colonoscopy Preparation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Full dose preparation; AM colonoscopy (Experimental): Four hourly doses of lactulose for oral solution are taken in the evening. The colonoscopy is initiated prior to noon on the following day.
  Interventions: Drug: Full dose preparation
- Full dose preparation; PM colonoscopy (Experimental): Four hourly doses of lactulose for oral solution are taken in the evening. The colonoscopy is initiated after noon on the following day.
  Interventions: Drug: Full dose preparation
- Split dose preparation; AM colonoscopy (Experimental): Three hourly doses of lactulose for oral solution are taken in the evening prior to the day of the colonoscopy procedure; one dose is taken on the morning of the procedure. The colonoscopy is initiated prior to noon.
  Interventions: Drug: Split dose preparation
- Split dose preparation; PM colonoscopy (Experimental): Three hourly doses of lactulose for oral solution are taken in the evening prior to the day of the colonoscopy procedure; one dose is taken on the morning of the procedure. The colonoscopy is initiated after noon.
  Interventions: Drug: Split dose preparation

INTERVENTIONS:
Drug: Full dose preparation
  Other Names: Evening-only Regimen
  Arms: Full dose preparation; AM colonoscopy; Full dose preparation; PM colonoscopy
Drug: Split dose preparation
  Arms: Split dose preparation; AM colonoscopy; Split dose preparation; PM colonoscopy

SUMMARY:
The purpose of the study is to determine the efficacy of 2 regimens of lactulose as a preparation for colonoscopy.

DETAILED DESCRIPTION:
A full-dose regimen of lactulose for oral solution, where all dosing is completed the evening prior to the colonoscopy procedure, will be studied and compared to a split-dose regimen, where three doses are taken on the prior evening, and one dose is taken the morning of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring bowel evacuation for colonoscopy.

Exclusion Criteria:

* Patients with galactosemia (galactose-sensitive diet).
* Patients known to be hypersensitive to any of the components of lactulose for oral solution.
* Patients with an abnormality on screening blood work or vital sign assessments that, in the Investigator's judgment, may pose a significant risk including those pertaining to dehydration or electrolyte shifts.
* Patients with a history of impaired renal function.
* Patients with current or recent history of hypotension, as defined by the Investigator.
* Patients with a history of long Q-T syndrome.
* Patients with a history of a failed bowel preparation.
* Patients with severe constipation, defined as those patients taking daily prescription or over-the-counter laxatives.
* Patients with possible bowel obstruction, gastric retention, bowel perforation, toxic colitis, toxic megacolon, ileus or previous colonic surgery.
* Patients on lactulose therapy or receiving any treatment for chronic constipation.
* Be pregnant or nursing.
* Patients with known large polyps or flat polyps (i.e. polyps requiring electrocautery or argon plasma coagulation).
* Patients less than 18 years of age.
* Inability to understand the requirements of the study or be unwilling to provide written informed consent (as evidenced by signature on an informed consent document approved by an Institutional Review Board [IRB]) and agree to abide by the study restrictions.
* Be otherwise unsuitable for the study, in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2013-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Krause, M.D, Principal Investigator — ClinSearch, LLC
Locations (1):
- ClinSearch, LLC, Chattanooga, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Full Dose Preparation; AM Colonoscopy: Four hourly doses of lactulose for oral solution are taken in the evening prior to the day of the colonoscopy procedure. The colonoscopy is initiated prior to noon.
- Full Dose Preparation; PM Colonoscopy: Four hourly doses of lactulose for oral solution are taken in the evening prior to the day of the colonoscopy procedure. The colonoscopy is initiated after noon.
Period: Overall Study
Arm/Group | Full Dose Preparation; AM Colonoscopy | Full Dose Preparation; PM Colonoscopy | Split Dose Preparation; AM Colonoscopy | Split Dose Preparation; PM Colonoscopy
Started | 10 | 10 | 10 | 10
Completed | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Full Dose Preparation: PM Colonoscopy: Four hourly doses of lactulose for oral solution are taken in the evening prior to the day of the colonoscopy procedure. The colonoscopy is initiated after noon.
- Split Dose Preparation; AM Colonscopy: Three hourly doses of lactulose for oral solution are taken in the evening prior to the day of the colonoscopy procedure; one dose is taken on the morning of the procedure. The colonoscopy is initiated prior to noon.
- Total: Total of all reporting groups
Arm/Group | Full Dose Preparation; AM Colonoscopy | Full Dose Preparation: PM Colonoscopy | Split Dose Preparation; AM Colonscopy | Split Dose Preparation; PM Colonoscopy | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 7 | 9 | 8 | 33
  >=65 years | 1 | 3 | 1 | 2 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 5 | 7 | 24
  Male | 4 | 4 | 5 | 3 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 10 | 10 | 10 | 9 | 39
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1
  White | 10 | 10 | 10 | 9 | 39
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Lactulose as a Preparation for Colonoscopy.
Description: Efficacy assessed by the physician's determination of the cleanliness of the colon using the cumulative Boston Bowel Preparation Scale (BBPS) score. The cumulative score is derived from three segmental scores assessed from the following three colonic segments: right colon, transverse colon, and left colon. Segment scores range from 0 to 3 with the following abbreviated definitions: 0=mucosa not visible; 1=a portion of the mucosa is visible; 2=minor residue, but mucosa is seen well; 3=entire mucosa is seen well with no residue.
  The cumulative BBPS score is the sum of the three segment scores such that a cumulative score of 9 represents a colon with maximum mucosa visible and a score of 0 represents minimal visibility.
Time Frame: at least 3 hours post last consumption
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Regimen A for AM Colonoscopy: Regimen A for morning colonoscopy
  Regimen A
- Regimen A for PM Colonoscopy: Regimen A for afternoon colonoscopy
  Regimen A
- Regimen B for AM Colonoscopy: Regimen B for morning colonoscopy
  Regimen B
- Regimen B for PM Colonoscopy: Regimen B for afternoon colonoscopy
  Regimen B
Arm/Group | Regimen A for AM Colonoscopy | Regimen A for PM Colonoscopy | Regimen B for AM Colonoscopy | Regimen B for PM Colonoscopy
Number analyzed (Participants) | 10 | 10 | 10 | 10
units on a scale | 8.2 (0.42) | 7.2 (1.23) | 7.5 (1.90) | 8.4 (1.26)

2. Secondary Outcome: Incidence of Treatment Failure
Description: A treatment failure is defined in the protocol as a bowel preparation that receives a cumulative Boston Bowel Preparation Score less than 5, or has one or more of the segments scored as a 0.
Time Frame: at least 3 hours post last consumption
Population: The study objectives in the protocol called for the incidence of treatment failures to be calculated from the pooled data of all treatment participants. Therefore, outcome measures are not displayed with respect to individual treatment groups.
Measure: Number; unit: participants
Groups:
- Lactulose for Oral Solution: All patients taking lactulose for oral solution.
Arm/Group | Lactulose for Oral Solution
Number analyzed (Participants) | 40
participants | 1

3. Secondary Outcome: Tolerability of and Preference for Lactulose as a Bowel Evacuant-Patient Visual Analog Scale (VAS)
Description: A paper questionnaire contained a horizontal line 100 mm long with the right end labeled "Best Possible Experience" and the left end labeled "Worst Possible Experience". The patients were asked to use a pen to place a mark on the line at the point that best described their overall tolerability for the bowel preparation.
  Scores were determined by measuring the distance of the mark from the left end of the line. So, a lower number would indicate a poor experience and a high number would reflect a positive experience, with 100 being the maximum score and one that describes the best possible experience with the preparation.
Time Frame: 3 - 15 hours post last consumption
Population: The study objectives in the protocol called for patient tolerability to be evaluated for all treatment participants. Therefore, outcome measures are not displayed with respect to the four individual treatment groups.
Measure: Mean (Standard Deviation); unit: units on VAS scale
Arm/Group | Lactulose for Oral Solution
Number analyzed (Participants) | 40
units on VAS scale | 79.6 (17.2)

4. Secondary Outcome: Tolerability of and Preference for Lactulose as a Bowel Evacuant-Likert 1
Description: Tolerability assessed by a patient questionnaire - Likert response to "was regimen a tolerable bowel prep?" Range of responses allowed include whole numbers between 1 and 7. The following guide was given to the patients: 1 = Strongly Disagree; 4 = Neutral; 7 = Strongly Agree
Time Frame: 3-15 hours post last consumption
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on Likert Scale
Arm/Group | Lactulose for Oral Solution
Number analyzed (Participants) | 40
units on Likert Scale | 6.0 (1.6)

5. Secondary Outcome: Tolerability of and Preference for Lactulose as a Bowel Evacuant-Likert 2
Description: Tolerability assessed by a patient questionnaire - Likert response to "I did not experience too much discomfort during the bowel prep" Range of responses allowed include whole numbers between 1 and 7. The following guide was given to the patients: 1 = Strongly Disagree; 4 = Neutral; 7 = Strongly Agree
Time Frame: 3-15 hours post last consumption
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on Likert Scale
Arm/Group | Lactulose for Oral Solution
Number analyzed (Participants) | 40
units on Likert Scale | 5.5 (2.1)

6. Secondary Outcome: Tolerability of and Preference for Lactulose as a Bowel Evacuant-Likert 3
Description: Tolerability assessed by a patient questionnaire - Likert response to "The dosing instructions were easy to understand and follow" Range of responses allowed include whole numbers between 1 and 7. The following guide was given to the patients: 1 = Strongly Disagree; 4 = Neutral; 7 = Strongly Agree
Time Frame: 3 - 15 hours post last consumption
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on Likert Scale
Groups:
- Lactulose for Oral Solution: All patients taking lactulose for oral solution
  .
Arm/Group | Lactulose for Oral Solution
Number analyzed (Participants) | 40
units on Likert Scale | 6.8 (0.9)

7. Secondary Outcome: Tolerability of and Preference for Lactulose as a Bowel Evacuant
Description: Survey response to question: "Would you be willing to repeat this preparation if a colonoscopy was felt to be medically necessary at some point in the future? The outcome measure is reporting the percentage of participants who replied "Yes" to this survey question.
Time Frame: 3 - 15 hours post last consumption
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Lactulose for Oral Solution
Number analyzed (Participants) | 40
Percentage of Participants | 93

8. Secondary Outcome: Tolerability of and Preference for Lactulose as a Bowel Evacuant
Description: Survey response to question: "if you had a previous colonoscopy, please indicate your preference for the crystalline lactulose or the previous medications.
Time Frame: 3 to 15 hours post last consumption
Population: Of the 40 participants responding to the patient questionnaire, only 21 reported that they had had a previous colonoscopy; therefore, the other 19 are not included in this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Lactulose for Oral Solution
Number analyzed (Participants) | 21
percentage of participants
  Strongly prefer the lactulose | 62
  Somewhat prefer the Lactulose | 24
  Have no preference | 5
  Somewhat prefer the other | 5
  Strongly prefer the other | 5

9. Secondary Outcome: Colonic Hydrogen Gas Levels
Time Frame: 3 - 15 hours post last consumption
Population: A secondary objective in the protocol called for colonic gas levels to be measured for all treatment participants. Therefore, outcome measures are not displayed with respect to the four individual treatment groups.
Measure: Mean (Standard Deviation); unit: parts per million by volume
Arm/Group | Lactulose for Oral Solution
Number analyzed (Participants) | 40
parts per million by volume
  Sigmoid colon; start of procedure | 1267 (3158)
  Cecum | 3637 (11297)
  Sigmoid colon; end procedure | 314 (329)

10. Secondary Outcome: Colonic Methane Gas Levels
Time Frame: 3 - 15 hours post last consumption
Population: as for outcome 9
Measure: Mean (Full Range); unit: parts per million by volume
Arm/Group | Lactulose for Oral Solution
Number analyzed (Participants) | 40
parts per million by volume | NA [NA to NA] — All values for methane were below the level of detection of the laboratory methods

ADVERSE EVENTS:
Time Frame: through one day following study drug consumption
Description: The safety endpoint defined in the protocol collected adverse events for all patients taking the investigational product. Comparisons between treatment groups were not intended according to the statistical plan and results are reported as one group.
Groups:
- Lactulose for Oral Solution: All patients taking lactulose for oral solution were evaluated as one group for purposes of providing survey data on the use of the product as a bowel preparation agent for colonoscopy.
Arm/Group | Lactulose for Oral Solution
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 7/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lactulose for Oral Solution (N=40)
Vomiting (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No